CLINICAL TRIAL: NCT00619216
Title: A Three-Month, Open-Label, Two Cohort Study to Investigate the Safety and Tolerability of Myfortic in Combination With Neoral (Cyclosporin) or Prograf (Tacrolimus) in Liver Transplant Recipients With GI Intolerance
Brief Title: Myfortic Conversion Trial in OLT Recipients With GI Intolerance
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: David Gerber, MD/Principal Investigator, UNC Department of Surgery
Other Study IDs: 07-1203
Record Dates: First submitted 2008-02-07; First posted 2008-02-20 (Estimated); Last update posted 2011-06-03 (Estimated); Status verified 2011-06

CONDITIONS: GI Disturbance
Keywords: Orthotopic Liver Transplant Recipients with GI disturbance
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Mycophenolic Acid (Myfortic) — Equimolar conversion from mycophenolate mofetil to mycophenolic acid
  Other Names: Cellcept; Myfortic

SUMMARY:
Liver transplant patients often require multimodal immunosuppressive therapy to minimize their risk for rejection. In our regimen, MMF (mycophenolate mofetil) is often added to lower the side effects of the calcineurin inhibitors. Unfortunately the literature reports 20% up to as many as 40% of patients have GI intolerance to MMF. At our Center, approximately 30% of patients have intolerance to MMF, thereby mitigating our ability to use this agent. The primary objective of this study is to assess the tolerability of myfortic in combination with Neoral or Tacrolimus as determined by the GSRS (Gastrointestinal Symptom Rating Scale) after conversion from MMF in maintenance liver transplant patients with GI intolerance within 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of orthotopic liver transplant at least 8 weeks post transplant
* Mild and/or moderate GI complaints directly related to MMF

Exclusion Criteria:

* Multi-organ transplant recipients
* Evidence of graft rejection within 14 days prior to Baseline visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recipients of Orthotopic Liver Transplants
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of GI symptoms using GSRS, GIQLi, and SF-12 after conversion to Myfortic | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: David Gerber, MD, Principal Investigator — UNC-Chapel Hill Department of Surgery
Locations (1):
- University of North Carolina-Chapel Hill, Chapel Hill, North Carolina, United States